CLINICAL TRIAL: NCT06064903
Title: Phase I/II Study of Anti-CD7 Chimeric Antigen Receptor-Expressing T Cells in Pediatric Patients Affected by Relapsed/Refractory CD7+ T-cell Acute Lymphoblastic Leukemia/Lymphoma
Brief Title: CD7-CAR-T Cells in Pediatric Relapsed/Refractory CD7+ T-ALL/LL
Acronym: CD7-CAR01
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD7-CAR01
Record Dates: First submitted 2023-09-12; First posted 2023-10-03 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: T-Cell Acute Lymphoblastic Leukemia/Lymphoblastic Lymphoma
Keywords: T-ALL; T-LL; Relapsed; Refractory; anti-CD7 PEBL-CAR T
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD7-CART01 (Experimental): A single IV infusion of CD7-CART01 (CD7-directed chimeric antigen receptor T-cells) on Day 0 after lymphodepleting regimen.
  Patients will receive the following lymphodepleting regimen:
  * Fludarabine 30 mg/m2 per day over 1 hour on days -6, -5, -4 and -3
  * Cyclophosphamide 1000 mg/m2 per day on days -4 and -3.
  CD7-CART01 will be infused at the following dose levels:
  * DL1: 0.5 x 10^6 CAR+ cells/kg
  * DL2: 1 x 10^6 CAR+ cells/kg
  If 2 DLTs are observed an additional DL0 of 0.25 x 106 CAR+ cells /kg will be explored.
  Interventions: Biological: CD7-CART01

INTERVENTIONS:
Biological: CD7-CART01 — A single IV infusion of CD7-CART01 on Day 0

SUMMARY:
The main purpose of this study is to evaluate the safety, to establish the recommended dose, and to evaluate the antitumor effect of CD7-CART01 in pediatric patients with relapsed or refractory (R/R) T-cell acute lymphoblastic leukemia (T-ALL) or lymphoblastic lymphoma (T-LL).

DETAILED DESCRIPTION:
This is an in-human, open-lable, single-arm, single-agent, Phase 1/2 study in pediatric patients with R/R T-ALL/T-LL who have failed at least one standard frontline chemotherapy or relapsed after allogeneic hematopoietic stem cell transplantation (HSCT). The study will consist of two phases, Phase 1 and Phase 2. During the Dose Escalation portion of the trial (Phase 1) up to 12 patients will receive CD7-CART01, in up to 2 dose levels until maximum tolerated dose (MTD) is determined. If 2 DLTs are observed in the dose level 1 an additional DL0 will be explored. The dose escalation phase will enroll successive cohorts of 3 up to 6 patients guided by a standard dose-finding 3 + 3 design. Once the recommended phase 2 dose (RP2D) is defined, the phase 2 portion of the study will enroll at the MTD/RD identified in the phase I up to 26 pediatric patients (for both phases) and the study protocol will be amended to include additional, international centers.

ELIGIBILITY:
Procurement eligibility

Inclusion Criteria:

1. Diagnosis of CD7 expressing (> 98% CD7 expression on blast cells) T-ALL or LL and one of the following:

   1. Patients in 1st or subsequent relapse, after at least one standard frontline chemotherapy with BM involvement (MRD >1% in 2 consecutive determinations or evidence of morphological relapse, i.e. >5% blasts in BM);
   2. Relapse after allogeneic HSCT, if at least 100 days post-transplant, if there is no evidence of active GVHD and if the patient is no longer taking immunosuppressive agents for at least 30 days prior to enrollment;
   3. CNS disease as defined as > 5 WBCs/mcL in CSF with morphological/flow-cytometry evidence of blasts or biopsy proven recurrence in the eye or brain;
   4. Extramedullary relapse as defined by morphological evidence of blasts in the testis or any other extramedullary sites;
   5. Refractory disease, defined as MRD ≥ 1% or <1% but persistently positive (i.e. a positive MRD value confirmed by PCR at 2 subsequent evaluations performed at least 2 weeks apart), at the end of consolidation blocks in newly diagnosed patients;
2. Age: 6 months - 25 years.
3. Adequate venous access for apheresis or eligible for appropriate catheter placement, and no other contraindications for leukapheresis.
4. Voluntary informed consent is given. For subjects <18-year-old, or below the age required by each Country regulation, their legal guardian must give informed consent. Pediatric subjects will be included in age-appropriate discussion and verbal assent will be obtained for those greater than or equal to 12 years of age, when appropriate, or to sign age-adapted informed consent, according to the regulatory requirement of each Country.
5. Clinical performance status: Patients > 16 years of age: Karnofsky greater than or equal to 60%; Patients < 16 years of age: Lansky scale greater than or equal to 60%.

Exclusion Criteria:

1. Severe, uncontrolled active intercurrent infections.
2. HIV, or active HCV and/or HBV infection.
3. Blast contamination in peripheral blood >5%, by flow-cytometry, at the time of leukapheresis collection.
4. Concurrent or recent prior therapies, before apheresis:

   1. Systemic steroids (at a dose equivalent to or greater than 2 mg/kg prednisone) in the 2 weeks before apheresis collection. Recent or current use of inhaled/topical/non-absorbable steroids is not exclusionary
   2. Systemic chemotherapy in the 2 weeks preceding apheresis collection
   3. Nelarabine, daratumomab, clofarabine exposure in the 3 weeks preceding apheresis collection
   4. Anti-thymocyte globulin (ATG) or Alemtuzumab (Campath®) in the 8 weeks preceding apheresis collection
   5. Immunosuppressive agents in the 2 weeks preceding apheresis collection
   6. Radiation therapy must have been completed at least 2 weeks prior to apheresis
   7. Other anti-neoplastic investigational agents currently administered or within 30 days prior to apheresis (i.e. start of protocol therapy)
   8. Exceptions:

      * There is no time restriction with regard to prior intrathecal chemotherapy, provided that there is complete recovery from any acute toxic effects of such chemotherapy;
      * Patients who relapse while receiving standard ALL maintenance chemotherapy will not be required to have a waiting period before entry onto this study provided they meet all other eligibility criteria;
      * Subjects receiving steroid therapy at physiologic replacement doses only are allowed provided there has been no increase in dose for at least 2 weeks prior to starting apheresis.

Treatment eligibility

Inclusion criteria:

1. Diagnosis of CD7 expressing (> 98% CD7 expression on blast cells) T-ALL or LL and one of the following:

   1. Patients in 1st or subsequent relapse, after at least one standard frontline chemotherapy with BM involvement (MRD >1% in 2 consecutive determinations or evidence of morphological relapse, i.e. >5% blasts in BM)
   2. Relapse after allogeneic HSCT, if at least 100 days post-transplant, if there is no evidence of active GVHD and if the patient is no longer taking immunosuppressive agents for at least 30 days prior to enrollment
   3. CNS disease as defined as > 5 WBCs/mcL in CSF with morphological or flow-cytometry evidence of blasts or biopsy proven recurrence in the eye or brain
   4. Extramedullary relapse as defined by morphological evidence of blasts in the testis or any other extramedullary sites
   5. Refractory disease, defined as MRD ≥1% or <1% but persistently positive (i.e. a positive MRD value confirmed by PCR at 2 subsequent evaluations performed at least 2 weeks apart), at the end of consolidation blocks in newly diagnosed patients
2. Measurable or evaluable disease at the time of enrollment, which may include any evidence of disease, including MRD detected by flow-cytometry, cytogenetics, or polymerase chain reaction (PCR) analysis.
3. Age: 6 months - 25 years.
4. Before enrollment for treatment, patients must have a potential allogeneic hematopoietic stem cell (HSC) donor (matched related, matched unrelated or haploidentical) available.
5. Voluntary informed consent is given. For subjects <18-year-old, or below the age required according to each Country regulation, their legal guardian must give informed consent. Pediatric subjects will be included in age-appropriate discussion and verbal assent will be obtained for those greater than or equal to 12 years of age, when appropriate, or to sign age-adapted informed consent, according to the regulatory requirement of the Country.
6. Clinical performance status: Patients > 16 years of age: Karnofsky greater than or equal to 60%; Patients < 16 years of age: Lansky scale greater than or equal to 60%.

Exclusion criteria:

1. Pregnant or lactating women.
2. Severe, uncontrolled active intercurrent infections.
3. HIV, or active HCV and/or HBV infection.
4. Life-expectancy < 6 weeks.
5. Hepatic function: Inadequate liver function defined as total bilirubin > 4x upper limit of normal (ULN) or transaminase (ALT and AST) > 6 x ULN.
6. Renal function: serum creatinine > 3x ULN for age.
7. Blood oxygen saturation < 90%.
8. Cardiac function: Left ventricular ejection fraction lower than 45% by ECHO.
9. Congestive heart failure, cardiac arrhythmia, psychiatric illness, or social situations that would limit compliance with study requirements or in the opinion of the PI would pose an unacceptable risk to the subject.
10. Uncontrolled seizures or status epilepticus; increased intra-cranial pressure as evidenced by papilledema and CSF opening pressure > 20 cm water; decreased conscious state (any cause).
11. Contamination of either the apheresis collection or the CD7-CART01 drug product with >5% blasts.
12. Presence of active, grade 2-4 acute or extensive chronic GvHD.
13. Concurrent or recent prior therapies, before infusion:

    1. Systemic steroids (at a dose > 2 mg/kg prednisone) in the 2 weeks before infusion. Recent or current use of inhaled/topical/non-absorbable steroids is not exclusionary
    2. Systemic chemotherapy in the 2 weeks preceding infusion
    3. Anti-thymocyte globulin (ATG) or Alemtuzumab (Campath®) in the 8 weeks preceding infusion
    4. Immunosuppressive agents in the 2 weeks preceding infusion
    5. Radiation therapy must have been completed at least 3 weeks prior to enrollment
    6. Other anti-neoplastic investigational agents currently administered or within 30 days prior to infusion (i.e., start of protocol therapy)
    7. Exceptions:

       * There is no time restriction in regards to prior intrathecal chemotherapy but there must be a complete recovery from any acute toxic effects from such chemotherapy;
       * Patients who relapse while receiving standard ALL maintenance chemotherapy will not be required to have a waiting period before entry onto this study provided that they meet all other eligibility criteria;
       * Subjects receiving steroid therapy at physiologic replacement doses only are allowed provided that there has been no increase in dose for at least 2 weeks prior to starting apheresis.

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-04-21 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2040-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety (Phase I) and definition of the recommended dose (Phase I) | 28 days
  To evaluate the safety of the infusion of CD7-CART01, explore the dose-limiting toxicities (DLT) of the cellular product and define the recommended dose of CD7-CART01, defined as the maximum tolerated dose/recommended dose (MTD/RD), to be evaluated for efficacy in the phase II extension
Antitumor effect of CD7-CART01 (Phase II) | 28 days
  To evaluate the portion of patients achieving either BM, PB and CSF morphological complete remission (CR) or CR with incomplete blood count recovery (CRi) and with minimal residual disease (MRD) negativity at day 28

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 28 days
  In the phase II portion of the study, the treatment-related adverse events will be recorded
Antitumor effect of CD7-CART01 (Phase I and II) | 28 days
  To assess the Overall Response Rate (ORR) at day 28
In vivo persistence of CD7-CART01 (Phase I and II) | 3 years
  To assess the in vivo persistence of the infused T cells using immunoassays and transgene detection (flow-cytometry and Real Time qPCR)
Relative proportion and phenotype of CD3+CAR+ T cells/CD3+CAR- T cells/NK cells (Phase I and II) | 3 years
  To assess the relative proportion and phenotype of CD3+CAR+ T cells/CD3+CAR- T cells/NK cells at day +28 and whenever it will be the case at subsequent time points
Assessment of cumulative incidence of relapse | 3 years
  To assess the cumulative incidence of both molecular and morphological relapse (defined as an MRD >10^-4 and a BM blast percentage > 5%, respectively)
Assessment of cumulative incidence of overall survival | 3 years
  To assess the cumulative incidence of overall survival at 1 and 3 years post cell infusion
Assessment of cumulative incidence of disease-free survival | 3 years
  To assess the cumulative incidence of disease-free survival at 1 and 3 years post cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Franco Locatelli, MD, PhD, Principal Investigator — Director Department of Hematology/Oncology and Cell and Gene Therapy
Locations (1):
- Ospedale Pediatrico Bambino Gesù, Rome, Rome, Italy